CLINICAL TRIAL: NCT01493778
Title: Safety and Efficacy of Turoctocog Alfa in Prevention and Treatment of Bleeds in Paediatric Previously Untreated Patients With Haemophilia A
Brief Title: Safety and Efficacy of Turoctocog Alfa in Prevention and Treatment of Bleeds in Previously Untreated Children With Haemophilia A
Acronym: guardian™4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7008-3809; U1111-1119-6116 (Other: WHO); 2011-001033-16 (EudraCT Number); P/50/2010 (Other: EMA (PDCO)); JapicCTI-142544 (Other: JAPIC); CTR20150455 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- turoctocog alfa (Experimental)
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Patients will be scheduled to receive treatment with turoctocog alfa for at least 100 exposure days. In most cases, treatment will be given at home with intravenous (i.v., into the vein) self-injection by the parent/caregiver/support person.

SUMMARY:
This trial is conducted in Asia, Europe and North America. The purpose of the trial is to evaluate the safety and efficacy of turoctocog alfa in prevention and treatment of bleeds in previously untreated children with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Age below 6 years
* Informed consent obtained before any trial-related activities (trial-related activities are any procedure that would not have been performed during normal management of the patient)
* Male patients diagnosed with congenital severe haemophilia A (FVIII level equal to or below 1%)
* No prior use of purified clotting factor products (previous exposure, equal to or less than 5 ED to blood components, e.g. cryoprecipitate, fresh frozen plasma, is accepted) including commercially available NovoEight® /Novoeight®

Exclusion Criteria:

* Known or suspected allergy to hamster protein or intolerance to trial product(s) or related products
* Previous participation in this trial defined as withdrawal after administration of trial product
* Congenital or acquired coagulation disorders other than haemophilia A
* Any history of Factor VIII inhibitor
* Ongoing treatment or planned treatment during the trial with immunomodulatory agents (e.g. intravenous immunoglobulin (IVIG), routine systemic corticosteroids)

Ages: 0 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (67):
- United States (23):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Macon, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Oak Lawn, Illinois
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, New Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Brooklyn, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
- Algeria (2):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Annaba
- Austria (7):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Innsbruck
  - Novo Nordisk Investigational Site, Klagenfurt
  - Novo Nordisk Investigational Site, Linz
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Sankt Pölten
  - Novo Nordisk Investigational Site, Vienna
- Brazil (2):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Campinas, São Paulo
- China (6):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chonqqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang
  - Novo Nordisk Investigational Site, Beijing
- Novo Nordisk Investigational Site, København Ø, Denmark
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Japan (4):
  - Novo Nordisk Investigational Site, Aichi
  - Novo Nordisk Investigational Site, Hyōgo
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Vilnius, Lithuania
- Poland (2):
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Lublin
- Novo Nordisk Investigational Site, Porto, Portugal
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (3):
  - Novo Nordisk Investigational Site, Krasnodar
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Spain (3):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, El Palmar
  - Novo Nordisk Investigational Site, Madrid
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, İzmit
  - Novo Nordisk Investigational Site, Samsun

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 40 sites in 15 countries: Algeria (1 site), Austria (2 sites), China (6 sites), Denmark (1 site), Greece (2 sites), Hong Kong (1 site), Hungary (1 site), Japan (2 sites), Lithuania (1 site), Poland (2 sites), Russian Federation (2 sites), Serbia (1 site), Spain (3 sites), Turkey (3 sites), United States (12).
Pre-assignment Details: Sixty (60) participants were enrolled in the trial and received at least one dose of turoctocog alfa.The trial consisted of two phases: the main phase including the screening visit (visit 1) and 4 subsequent visits, and an extension phase with a rolling visit schedule consisting of 6 planned visits including 4 dispensing visits) per year.
Groups:
- Turoctocog Alfa (N8) (Preventive+On-demand Treatment): Participants received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. Participants who enrolled into the trial initiated the preventive treatment no later than their second birthday or after a maximum of 2 bleeding episodes requiring treatment, whichever came first. The trial consisted of two phases. In the main phase, an aggregated number of at least 50 participants received preventive treatment with turoctocog alfa until they reached a minimum of 50 exposure days (ED) or until they developed inhibitors. After that the participants continued in the extension phase where at least 50 participants achieved at least 100 ED, which translated into a maximum trial duration of up to 5 years (including any potential inhibitor treatment). The estimated total duration of the trial was approximately 7 years.
Period: Overall Study
Arm/Group | Turoctocog Alfa (N8) (Preventive+On-demand Treatment)
Started | 60
Completed | 52
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all dosed participants with data after dosing.
Groups:
- Turoctocog Alfa (N8) (Preventive+On-demand): Participants received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. Participants who enrolled into the trial initiated the preventive treatment no later than their second birthday or after a maximum of 2 bleeding episodes requiring treatment, whichever came first. The trial consisted of two phases. In the main phase, an aggregated number of at least 50 participants received preventive treatment with turoctocog alfa until they reached a minimum of 50 exposure days (ED) or until they developed inhibitors. After that the participants continued in the extension phase where at least 50 participants achieved at least 100 ED, which translated into a maximum trial duration of up to 5 years (including any potential inhibitor treatment). The estimated total duration of the trial was approximately 7 years.
Arm/Group | Turoctocog Alfa (N8) (Preventive+On-demand)
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.2 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 44
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Factor VIII Inhibitors (Above or Equal to 0.6 BU (Bethesda Units)/mL) for the Main Phase of the Trial
Description: The incidence rate (percentage of participants with inhibitors) of inhibitors defined as inhibitor titres ≥0.6 BU for main phase of the trial.
Time Frame: From Visit 2 (21 days after screening) to Visit 5 (50-55 exposure day)
Population: Analysis was based on participants who completed the main phase of the trial.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Turoctocog Alfa (N8): Main Phase (Preventive Treatment): Participants received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. Subjects received prophylactic factor VIII replacement therapy (preventive treatment) until Visit 5 or until development of inhibitor, whichever came first. In the main phase, an aggregated number of at least 50 participants received preventive treatment with turoctocog alfa until they reached a minimum of 50 exposure days (ED) or until they developed inhibitors.
Arm/Group | Turoctocog Alfa (N8): Main Phase (Preventive Treatment)
Number analyzed (Participants) | 58
Percentage of participants | 43.1 [30.2 to 56.8]

2. Secondary Outcome: Haemostatic Effect of Turoctocog Alfa on Treatment of Bleeds Assessed on a Predefined Four Point Scale: Excellent, Good, Moderate and None
Description: The haemostatic effect of turoctocog alfa was summarised by frequency tables containing count of all bleeds and assessed on a predefined four point scale: Excellent, Good, Moderate and None. The analysis was based on the total number of bleeds and their response to treatment. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: From Visit 2 to Visit 5 (50-55 exposure day); From Visit 6 to end of trial, extension phase of the trial; From Visit 2 to end of trial, the combined main and extension phases of the trial
Population: The full analysis set included all dosed participants with data after dosing.
Measure: Count of Units; unit: bleeds
Units Other Than Participants: bleeds
Groups:
- Turoctocog Alfa (N8): Main Phase (On-demand Treatment): Participants (children≤2 years) received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection as on-demand treatment while waiting to start on a preventive regimen. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. This treatment period included Visit 2 to first preventive dose.
- Turoctocog Alfa (N8): Extension Phase (Preventive Treatment): Participants received prophylactic treatment administered from completion of the main phase or completion of the inhibitor cohort until the end-of-trial visit in the extension phase. They received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. After completing the main phase, participants continued in the extension phase where at least 50 participants achieved at least 100 ED, which translated into a maximum trial duration of up to 5 years (including any potential inhibitor treatment).
- Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment: Participants who started preventive treatment in the main and extension phase are included in this arm. They received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the child's clinical profile. The trial consisted of two phases. In the main phase, an aggregated number of at least 50 participants received preventive treatment with turoctocog alfa until they reached a minimum of 50 exposure days (ED) or until they developed inhibitors. After that the participants continued in the extension phase where at least 50 participants achieved at least 100 ED, which translated into a maximum trial duration of up to 5 years (including any potential inhibitor treatment). The estimated total duration of the trial was approximately 7 years.
- Turoctocog Alfa (N8): Inhibitor Cohort: Participants who developed an inhibitor during the course of the trial and followed an alternative treatment regimen are included in this arm. They were offered continued treatment with turoctocog alfa for up to 24 months.
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
Number analyzed (bleeds) | 98 | 133 | 269 | 402 | 179
bleeds
  Excellent | 53 | 83 | 161 | 244 | 9
  Good | 36 | 29 | 73 | 102 | 19
  Moderate | 5 | 12 | 31 | 43 | 10
  None | 0 | 1 | 1 | 2 | 4
  Missing | 4 | 8 | 3 | 11 | 137

3. Secondary Outcome: Annualised Bleeding Rate (ABR)
Description: Annualised bleeding rate defined as number of bleeds in total per patient per year following treatment were estimated by a Poisson model allowing for over-dispersion. The Poisson estimate is presented with a 95% confidence interval (CI). The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: The full analysis (FAS) set included all dosed participants with data after dosing. Participants in FAS with only one exposure day were excluded from preventive treatment in main when calculating the Poisson estimates of ABR as the small amount of information introduces uncertainty to the estimated ABR.
Measure: Mean (95% Confidence Interval); unit: bleeds/patient/year
Units Other Than Participants: bleeding episodes
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
Number analyzed (bleeding episodes) | 98 | 133 | 269 | 402 | 179
bleeds/patient/year | 4.27 [3.09 to 5.89] | 5.63 [4.27 to 7.43] | 3.81 [2.84 to 5.11] | 4.26 [3.34 to 5.44] | 6.09 [3.77 to 9.84]

4. Secondary Outcome: Number of Turoctocog Alfa (N8) Injections Required Per Bleed
Description: The number of injections of turoctocog alfa (N8) required per bleed was calculated as the number of injections of turoctocog alfa used in the time period from start of the bleed to stop of the bleed. The mean number of turoctocog alfa injections required to stop the bleed is presented. The analysis was based on the total number of bleeds. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: Full Analysis Set included all dosed participants with data after dosing. Number of participants analysed=number of participants with bleeding episodes.
Measure: Mean (Standard Deviation); unit: injections/bleed
Units Other Than Participants: bleeds
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 36 | 38 | 40 | 52 | 26
Number analyzed (bleeds) | 98 | 133 | 269 | 402 | 179
injections/bleed | 2.1 (2.18) | 1.8 (2.98) | 2.4 (3.04) | 2.2 (3.03) | 2.8 (6.24)

5. Secondary Outcome: Total Consumption of Turoctocog Alfa (N8) Per Patient (Prevention, Treatment of Bleeds and During Surgery) Per Month
Description: Mean total consumption of turoctocog alfa (N8) used for treatment (includes all injections given: prevention, treatment of bleeds and during surgery) per patient per month. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: Full Analysis Set included all dosed participants with data after dosing.
Measure: Mean (Standard Deviation); unit: IU/kg/month/patient
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
IU/kg/month/patient | 117.6 (190.7) | 359.8 (323.2) | 476.9 (209.3) | 437.2 (244.4) | 1815.2 (1653.8)

6. Secondary Outcome: Total Consumption of Turoctocog Alfa (N8) Per Patient (Prevention, Treatment of Bleeds and During Surgery) Per Year
Description: Mean total consumption of turoctocog alfa (N8) used for treatment (includes all injections given: prevention, treatment of bleeds and during surgery) per patient per year. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: Full Analysis Set included all dosed participants with data after dosing.
Measure: Mean (Standard Deviation); unit: IU/kg/year/patient
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
IU/kg/year/patient | 1410.8 (2288.4) | 4317.2 (3878.9) | 5722.5 (2512.0) | 5245.9 (2933.1) | 21782.8 (19845.6)

7. Secondary Outcome: Consumption of Turoctocog Alfa (N8) (IU/kg/Bleed) Per Bleed
Description: Mean consumption of turoctocog alfa (N8) used for treatment of bleed from start to stop of bleed. The analysis was based on number of bleeds. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: The full analysis set included all dosed participants with data after dosing.
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Units Other Than Participants: bleeds
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
Number analyzed (bleeds) | 98 | 133 | 269 | 402 | 179
IU/kg/bleed | 86.1 (116.8) | 80.8 (126.4) | 107.9 (137.7) | 98.9 (134.5) | 279.1 (821.7)

8. Secondary Outcome: Consumption of Turoctocog Alfa (N8) (IU/kg/Months) for Bleed Prevention
Description: Mean consumption of turoctocog alfa (N8) used for preventive treatment per month per patient. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: The full analysis set included all dosed participants with data after dosing. Participants in on-demand treatment did not receive treatment for bleed prevention and therefore are not included in the analysis.
Measure: Mean (Standard Deviation); unit: IU/kg/month/patient
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 0 | 58 | 49 | 59 | 26
IU/kg/month/patient |  | 293.5 (281.1) | 446.3 (206.2) | 399.0 (234.7) | 1692.6 (1553.9)

9. Secondary Outcome: Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) Reported During the Trial Period
Description: Number of adverse events and serious adverse events per patient years of exposure. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial (exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: The safety analysis set included all dosed participants with data after dosing. The arm group - 'main phase' includes subjects who were treated both on-demand and preventively in the main phase. 'On-Demand' and 'Preventive' were not described as separate arms/groups in the protocol. These were not analysed separately for this endpoint.
Measure: Number; unit: events per patient years of exposure
Arm/Group | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 60 | 49 | 60 | 26
events per patient years of exposure
  All adverse events | 5.85 | 3.76 | 5.12 | 7.41
  Serious adverse events | 1.02 | 0.24 | 0.73 | 1.52

10. Secondary Outcome: Incidence Rate of Clinically Relevant Inhibitors Defined as an Inhibitor Titre (≥ 0.6 BU/mL) Combined With a Decreased Recovery (<66% of Expected Level)
Description: The incidence rates (number of patients with new inhibitor in the period/number of participants at risk, expressed in percentage) of clinically relevant inhibitors were defined as an inhibitor titre (≥ 0.6 BU) combined with a decreased recovery (<66% of expected level). Incidence rate of clinically relevant inhibitors according to the type of assay used is presented. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation) and the combined main and extension phase (from Visit 2 to end of trial).
Time Frame: as for outcome 2
Population: The full analysis set included all dosed participants with data after dosing. The arm group - 'main phase' includes subjects who were treated both on-demand and preventively in the main phase. 'On-Demand' and 'Preventive' were not described as separate arms/groups in the protocol. These were not analysed separately for this endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment
Number analyzed (Participants) | 58 | 33 | 58
Percentage of participants
  One-stage FVIII clotting activity assay | 36.2 [24.0 to 49.9] | 3.0 [0.1 to 15.8] | 37.9 [25.5 to 51.6]
  Two-stage chromogenic assay | 36.2 [24.0 to 49.9] | 3.0 [0.1 to 15.8] | 37.9 [25.5 to 51.6]

11. Secondary Outcome: Incidence Rate of High-titre Inhibitors Defined as Inhibitor Titre ≥ 5 BU (Bethesda Units)/mL)
Description: Incidence rate (number of patients with new inhibitor in the period/number of participants at risk, expressed in percentage) of high-titre inhibitors defined as inhibitor titre ≥ 5 BU (Bethesda Units)/mL). The inhibitors were evaluated for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation) and the combined main and extension phase (from Visit 2 to end of trial).
Time Frame: as for outcome 2
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment
Number analyzed (Participants) | 58 | 33 | 58
Percentage of participants | 27.6 [16.7 to 40.9] | 0.0 [0.0 to 10.6] | 27.6 [16.7 to 40.9]

12. Secondary Outcome: Change in Total Scores for Parent Reported Treatment Satisfaction
Description: The caregivers/parent reported treatment satisfaction is assessed by the parents using the haemophilia satisfaction questionnaire (HEMO-SAT). The questionnaire contained questions related to treatment that covered 6 domains (ease and convenience, efficacy, burden, specialist, centre and general satisfaction). Adults completing the questionnaire could achieve a score from 0 to 100, with lower scores reflecting greater treatment satisfaction. The scale range for each of the 6 domains was 0-100 with lower scores reflecting greater treatment satisfaction.
  The scores of the domains at visit 3 (10th-15th ED), visit 5 (50th-55th ED) and end of trial (EoT) are presented.
Time Frame: Visit 3 (10th-15th ED); Visit 5 (50th-55th ED); End of trial (within 8 weeks of their last scheduled visit in the extension phase)
Population: The full analysis set included all dosed participants with data after dosing. Number of participants analysed=number of participants who answered the questionnaire
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment
Number analyzed (Participants) | 59
Score on a scale
  Ease/convenience visit 3 Range: 0 - 100: number analyzed (Participants) | 36
  Ease/convenience visit 3 Range: 0 - 100 | 27.1 (14.6)
  Ease and convenience - visit 5 Score range: 0-100: number analyzed (Participants) | 26
  Ease and convenience - visit 5 Score range: 0-100 | 21.4 (14.9)
  Ease and convenience - EoT Score range:0-100: number analyzed (Participants) | 43
  Ease and convenience - EoT Score range:0-100 | 21.9 (13.4)
  Efficacy - visit 3 Score range: 0-100: number analyzed (Participants) | 36
  Efficacy - visit 3 Score range: 0-100 | 10.2 (12.8)
  Efficacy - visit 5 Score range: 0-100: number analyzed (Participants) | 26
  Efficacy - visit 5 Score range: 0-100 | 9.8 (10.5)
  Efficacy - end of trial Score range: 0-100: number analyzed (Participants) | 43
  Efficacy - end of trial Score range: 0-100 | 11.7 (17.4)
  Burden - visit 3 Score range: 0-100: number analyzed (Participants) | 35
  Burden - visit 3 Score range: 0-100 | 20.5 (21.0)
  Burden - visit 5 Score range: 0-100: number analyzed (Participants) | 26
  Burden - visit 5 Score range: 0-100 | 15.4 (17.4)
  Burden - end of trial Score range: 0-100: number analyzed (Participants) | 43
  Burden - end of trial Score range: 0-100 | 16.9 (16.6)
  Specialist/Nurses- visit 3 Score range: 0-100: number analyzed (Participants) | 37
  Specialist/Nurses- visit 3 Score range: 0-100 | 4.1 (8.4)
  Specialist/Nurses- visit 5 Score range: 0-100: number analyzed (Participants) | 26
  Specialist/Nurses- visit 5 Score range: 0-100 | 4.0 (6.6)
  Specialist/Nurses- end of trial Score range: 0-100: number analyzed (Participants) | 43
  Specialist/Nurses- end of trial Score range: 0-100 | 4.9 (8.2)
  Centre/Hospital - visit 3 Score range: 0-100: number analyzed (Participants) | 37
  Centre/Hospital - visit 3 Score range: 0-100 | 2.8 (5.7)
  Centre/Hospital - visit 5 Score range: 0-100: number analyzed (Participants) | 26
  Centre/Hospital - visit 5 Score range: 0-100 | 3.1 (5.7)
  Centre/Hospital - end of trial Score range: 0-100: number analyzed (Participants) | 43
  Centre/Hospital - end of trial Score range: 0-100 | 5.0 (8.9)
  General satisfaction - visit 3 Score range: 0-100: number analyzed (Participants) | 35
  General satisfaction - visit 3 Score range: 0-100 | 5.7 (10.7)
  General satisfaction - visit 5 Score range: 0-100: number analyzed (Participants) | 26
  General satisfaction - visit 5 Score range: 0-100 | 3.8 (8.5)
  General satisfaction - end of trial Range: 0-100: number analyzed (Participants) | 43
  General satisfaction - end of trial Range: 0-100 | 6.4 (15.3)

13. Secondary Outcome: Health Resource Utilization and Caregiver Burden Associated With Bleeds (Per Month Per Patient)
Description: Resource utilisation and caregiver burden are analysed in terms of average number of days absent from work and use of mobility aids (e.g. wheelchair or crutches) as a consequence of bleeds. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: The full analysis set included all dosed participants with data after dosing. Number of participants analysed=number of participants with data available
Measure: Mean (Standard Deviation); unit: days/month/patient
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
days/month/patient
  Caregiver/parent's absence from work: number analyzed (Participants) | 41 | 49 | 41 | 51 | 24
  Caregiver/parent's absence from work | 0.011 (0.050) | 0.533 (1.645) | 0.007 (0.027) | 0.232 (1.117) | 0.271 (0.641)
  Patient's use of mobility aids: number analyzed (Participants) | 40 | 48 | 41 | 51 | 24
  Patient's use of mobility aids | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.025 (0.084)

14. Secondary Outcome: Health Resource Utilization and Caregiver Burden Associated With Bleeds (Per Year Per Patient)
Description: Resource utilisation and caregiver burden are analysed in terms of average number of days of absence from work and use of mobility aids (e.g. wheelchair or crutches) as a consequence of bleeds. The analysis was performed for the main phase (from Visit 2 to Visit 5 [50-55 exposure day], extension phase (from Visit 6 to end of trial; exposure day 100, expected to occur between 6 and 48 months of trial participation), the combined main and extension phase (from Visit 2 to end of trial) and for the inhibitor cohort.
Time Frame: as for outcome 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days/year/patient
Arm/Group | Turoctocog Alfa (N8): Main Phase (On-demand Treatment) | Turoctocog Alfa (N8): Main Phase (Preventive Treatment) | Turoctocog Alfa (N8): Extension Phase (Preventive Treatment) | Turoctocog Alfa (N8): Combined-Main+Ext, Preventive Treatment | Turoctocog Alfa (N8): Inhibitor Cohort
Number analyzed (Participants) | 51 | 58 | 49 | 59 | 26
days/year/patient
  Caregiver/parent's absence from work: number analyzed (Participants) | 41 | 49 | 41 | 51 | 24
  Caregiver/parent's absence from work | 0.127 (0.601) | 6.396 (19.736) | 0.082 (0.319) | 2.779 (13.406) | 3.252 (7.691)
  Patient's use of mobility aids: number analyzed (Participants) | 40 | 48 | 41 | 51 | 24
  Patient's use of mobility aids | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.296 (1.006)

ADVERSE EVENTS:
Time Frame: Adverse events from the first trial related activity after the participant had signed the informed consent (visit 1) until the end-of-trial visit (within 8 weeks of their last scheduled visit in the extension phase; 100th exposure day).
Description: Reported adverse events were based on the safety analysis set including all dosed participants with data after dosing.
Groups:
- Turoctocog Alfa: Participants received turoctocog alfa doses of 15-60 IU/kg body weight (BW) administered as an intravenous injection for the prevention of bleeding. The investigator decided what dose of turoctocog alfa to give based on the participant's clinical profile. Participants who enrolled into the trial initiated the preventive treatment no later than their second birthday or after a maximum of 2 bleeding episodes requiring treatment, whichever came first. The trial consists of two phases. In the main phase, an aggregated number of at least 50 participants received preventive treatment with turoctocog alfa until they reach a minimum of 50 exposure days (ED) or until they developed inhibitors. After that the participants continued in the extension phase where at least 50 participants achieved at least 100 ED, which will translate into a maximum trial duration of up to 5 years (including any potential inhibitor treatment). The estimated total duration of the trial was approximately 7 years.
Arm/Group | Turoctocog Alfa
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 36/60
Other Adverse Events (participants affected / at risk) | 55/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turoctocog Alfa (N=60)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Catheter site haematoma (General disorders) | 2 (2)
Catheter site infection (Infections and infestations) | 2 (6)
Catheter site oedema (General disorders) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (2)
Central venous catheterisation (Surgical and medical procedures) | 2 (2)
Circumcision (Surgical and medical procedures) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1)
Device damage (Product Issues) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device related infection (Infections and infestations) | 3 (5)
Drug hypersensitivity (Immune system disorders) | 2 (2)
Factor VIII inhibition (Blood and lymphatic system disorders) | 25 (27)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Phlebitis deep (Vascular disorders) | 1 (1)
Poor venous access (Vascular disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Respiratory tract infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (3)
Staphylococcal infection (Infections and infestations) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Systemic bacterial infection (Infections and infestations) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Vascular device infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turoctocog Alfa (N=60)
Anaemia (Blood and lymphatic system disorders) | 6 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 4 (5)
Balanoposthitis (Reproductive system and breast disorders) | 3 (3)
Body temperature increased (Investigations) | 3 (4)
Bronchitis (Infections and infestations) | 7 (7)
Catheter site infection (Infections and infestations) | 3 (7)
Catheter site inflammation (General disorders) | 3 (3)
Conjunctivitis (Infections and infestations) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (26)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 12 (25)
Ear infection (Infections and infestations) | 6 (10)
Eczema (Skin and subcutaneous tissue disorders) | 5 (6)
Factor VIII inhibition (Blood and lymphatic system disorders) | 4 (4)
Gastroenteritis (Infections and infestations) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 3 (4)
Hand-foot-and-mouth disease (Infections and infestations) | 4 (5)
Head injury (Injury, poisoning and procedural complications) | 5 (9)
Influenza (Infections and infestations) | 5 (5)
Iron deficiency (Metabolism and nutrition disorders) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nasopharyngitis (Infections and infestations) | 16 (36)
Otitis media (Infections and infestations) | 4 (4)
Otitis media acute (Infections and infestations) | 4 (7)
Pharyngitis (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 5 (5)
Pyrexia (General disorders) | 32 (85)
Rash (Skin and subcutaneous tissue disorders) | 5 (11)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Teething (Gastrointestinal disorders) | 3 (3)
Tonsillitis (Infections and infestations) | 3 (6)
Upper respiratory tract infection (Infections and infestations) | 15 (64)
Varicella (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 7 (9)
Viral upper respiratory tract infection (Infections and infestations) | 4 (11)
Vomiting (Gastrointestinal disorders) | 11 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT01493778/Prot_SAP_000.pdf